CLINICAL TRIAL: NCT02090855
Title: A Re-Read Study to Compare the Brain Uptake of [18F]Flutemetamol With Brain Neuritic Plaque Density Determined Postmortem.
Brief Title: Re-Read Study to Compare the Brain Uptake of [18F]Flutemetamol With Brain Neuritic Plaque Density Determined Postmortem
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Covance (Industry); H2O Clinical LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-067-026
Record Dates: First submitted 2014-03-11; First posted 2014-03-18 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Brain specimen retained. Subjects who had previously been dosed with Flutemetamol (18F) Injection and imaged in Study GE067-007.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Flutemetamol (18F): There are no interventions in this study. This study is to assess the images taken previously from another study, GE-067-007.

SUMMARY:
Data from subjects who had previously been dosed with Flutemetamol (18F) Injection and imaged in Study GE-067-007, and who died on or before 10 June 2013, will be analyzed. The PET brain images previously obtained in Study GE-067-007 will be interpreted visually in randomized by 5 independent readers who are blinded to all other subject information, and the images will be classified as abnormal (positive for abnormal neuritic plaque density) or normal (negative for abnormal neuritic plaque density). The numbers of images in each category will be used to calculate sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* The subject was enrolled in prior Study GE067-007.
* The subject died on or before 10 June 2013.
* The subject's brain is judged to be of suitable quality for analysis, including all regions necessary for analysis.

Exclusion Criteria:

* Not Applicable

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who had previously been dosed with Flutemetamol (18F) Injection and imaged in Study GE067-007.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, M.D., Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Kim SJ, Jang H, Yoo H, Na DL, Ham H, Kim HJ, Kim JP, Farrar G, Moon SH, Seo SW. Clinical and Pathological Validation of CT-Based Regional Harmonization Methods of Amyloid PET. Clin Nucl Med. 2024 Jan 1;49(1):1-8. doi: 10.1097/RLU.0000000000004937. Epub 2023 Nov 29. PMID 38048354
- [Derived] Tome SO, Tsaka G, Ronisz A, Ospitalieri S, Gawor K, Gomes LA, Otto M, von Arnim CAF, Van Damme P, Van Den Bosch L, Ghebremedhin E, Laureyssen C, Sleegers K, Vandenberghe R, Rousseau F, Schymkowitz J, Thal DR. TDP-43 pathology is associated with increased tau burdens and seeding. Mol Neurodegener. 2023 Sep 30;18(1):71. doi: 10.1186/s13024-023-00653-0. PMID 37777806
- [Derived] Thal DR, Ronisz A, Tousseyn T, Rijal Upadhaya A, Balakrishnan K, Vandenberghe R, Vandenbulcke M, von Arnim CAF, Otto M, Beach TG, Lilja J, Heurling K, Chakrabarty A, Ismail A, Buckley C, Smith APL, Kumar S, Farrar G, Walter J. Different aspects of Alzheimer's disease-related amyloid beta-peptide pathology and their relationship to amyloid positron emission tomography imaging and dementia. Acta Neuropathol Commun. 2019 Nov 14;7(1):178. doi: 10.1186/s40478-019-0837-9. PMID 31727169
- [Derived] Thal DR, Beach TG, Zanette M, Lilja J, Heurling K, Chakrabarty A, Ismail A, Farrar G, Buckley C, Smith APL. Estimation of amyloid distribution by [18F]flutemetamol PET predicts the neuropathological phase of amyloid beta-protein deposition. Acta Neuropathol. 2018 Oct;136(4):557-567. doi: 10.1007/s00401-018-1897-9. Epub 2018 Aug 19. PMID 30123935
- [Derived] Ikonomovic MD, Buckley CJ, Heurling K, Sherwin P, Jones PA, Zanette M, Mathis CA, Klunk WE, Chakrabarty A, Ironside J, Ismail A, Smith C, Thal DR, Beach TG, Farrar G, Smith AP. Post-mortem histopathology underlying beta-amyloid PET imaging following flutemetamol F 18 injection. Acta Neuropathol Commun. 2016 Dec 12;4(1):130. doi: 10.1186/s40478-016-0399-z. PMID 27955679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is to assess the images taken previously from another study, GE-067-007. No drug was administered. Subjects were previously dosed in Study GE-067-007.
Groups:
- Flutemetamol (18F): There are no interventions in this study. This study is to assess the images taken previously from another study, GE-067-007. No drug was administered. Subjects were previously dosed in Study GE-067-007.
Period: Overall Study
Arm/Group | Flutemetamol (18F)
Started | 108
Completed | 106
Not Completed | 2
Not completed — no evaluable Standard of Truth results | 2

BASELINE CHARACTERISTICS:
Population: This study is to assess the images taken previously from another study, GE-067-007. No drug was administered.
Groups:
- Flutemetamol (18F): There are no interventions in this study. This study is to assess the images taken previously from another study, GE-067-007. No drug was administered.
Arm/Group | Flutemetamol (18F)
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.8 (8.87)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 102
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: The Number of Abnormal Blinded Visual PET Image Interpretations.
Description: Blinded visual assessment of each subject's Flutemetamol (18F) Injection brain PET images as positive or negative will be performed by 5 independent blinded readers trained in the interpretation of [18F]flutemetamol PET images through an electronic training program.
Time Frame: Brain images will be assessed up to 1 year post subject's death.
Population: There are 76 autopsy cases confirmed to be abnormal. The majority interpretation is the interpretation made independently by more than half of the readers.
Measure: Number; unit: Number of Blinded Image Interpretations
Groups:
- Standard of Truth (SoT): Each Reader will have a total of 76 image interpretations when combining normal and abnormal readings.The Standard of Truth is based on moderate/frequent neuritic (amyloid) plaques, per modified Consortium to Establish a Registry for Alzheimer's Disease (CERAD) criteria, based on specimens stained with the Bielschowsky silver stain.
Arm/Group | Standard of Truth (SoT)
Number analyzed (Participants) | 76
Number of Blinded Image Interpretations
  Reader 1-Blinded Visual--Abnormal Interpretation | 73 [88.9 to 99.2]
  Reader 2-Blinded Visual--Abnormal Interpretation | 68 [80.3 to 95.3]
  Reader 3-Blinded Visual--Abnormal Interpretation | 67 [78.7 to 94.4]
  Reader 4-Blinded Visual--Abnormal Interpretation | 67 [78.7 to 94.4]
  Reader 5-Blinded Visual--Abnormal Interpretation | 72 [87.1 to 98.5]
  Majority Read-Abnormal | 69 [81.9 to 96.2]

2. Secondary Outcome: Number of Blinded Visual PET Image Interpretations
Description: Specificity of blinded visual image interpretations according to neuropathological criteria.
Time Frame: Brain images will be assessed up to 1 year post subject's death.
Population: There are 30 autopsy cases confirmed to be normal. The majority interpretation is the interpretation made independently by more than half of the readers.
Measure: Number; unit: Number of Blinded Image Intrepretations
Groups:
- Standard of Truth (SoT): Each Reader will have a total of 30 image interpretations when combining normal and abnormal readings.The Standard of Truth (SoT) is based on no/sparse neuritic (amyloid) plaques, per modified Consortium to Establish a Registry for Alzheimer's Disease (CERAD) criteria based on specimens stained with the Bielschowsky silver stain.
Arm/Group | Standard of Truth (SoT)
Number analyzed (Participants) | 30
Number of Blinded Image Intrepretations
  Reader 1-Blinded Visual-Normal Interpretation | 25
  Reader 2-Blinded Visual-Normal Interpretation | 27
  Reader 3-Blinded Visual-Normal Interpretation | 28
  Reader 4-Blinded Visual-Normal Interpretation | 25
  Reader 5-Blinded Visual-Normal Interpretation | 26
  Majority Read-Normal | 27

3. Primary Outcome: Sensitivity Percentage of Blinded Visual PET Image Interpretations of Subjects With Abnormal Scans
Description: as for outcome 1
Time Frame: Brain images will be assessed up to 1 year post subject's death.
Population: as for outcome 1
Measure: Number; unit: Percent of Sensitivity
Groups:
- Percentage of Sensitivity With Abnormal Reads: This is the percent of sensitivity with the Abnormal image interpretations.
Arm/Group | Percentage of Sensitivity With Abnormal Reads
Number analyzed (Participants) | 76
Percent of Sensitivity
  Reader 1-Blinded Visual--Abnormal Interpretation | 96.1
  Reader 2-Blinded Visual--Abnormal Interpretation | 89.5
  Reader 3-Blinded Visual--Abnormal Interpretation | 88.2
  Reader 4-Blinded Visual--Abnormal Interpretation | 88.2
  Reader 5-Blinded Visual--Abnormal Interpretation | 94.7
  Majority Read-Abnormal | 90.8

4. Secondary Outcome: Specificity Percentage of Blinded Visual PET Image Interpretations
Description: Specificity of blinded visual image interpretations according to neuropathological criteria, which is defined as the neuritic plaque density, neurofibriilary tangles and vasculpoathy in the brain.
Time Frame: Brain images will be assessed up to 1 year post subject's death.
Population: as for outcome 2
Measure: Number; unit: Percentage of Specificity
Groups:
- Percentage of Specificity for Normal Reads: This is the percentage of Specificity with the normal image interpretations.
Arm/Group | Percentage of Specificity for Normal Reads
Number analyzed (Participants) | 30
Percentage of Specificity
  Reader 1-Blinded Visual-Normal Interpretation | 83.3
  Reader 2-Blinded Visual-Normal Interpretation | 90.0
  Reader 3-Blinded Visual-Normal Interpretation | 93.3
  Reader 4-Blinded Visual-Normal Interpretation | 83.3
  Reader 5-Blinded Visual-Normal Interpretation | 86.7
  Majority Read-Normal | 90.0

ADVERSE EVENTS:
Description: Adverse events were not assessed nor collected in this study. In addition, no drug was administered. Therefore, this study had no adverse events. Subjects were previously dosed in Study GE-067-007.
Groups:
- Flutemetamol (18F): This study was to assess the PET images only. There was no drug administered in this study.
Arm/Group | Flutemetamol (18F)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The Clinical Trials NCT number is 01165554 for GE Healthcare study, GE-067-007.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No